CLINICAL TRIAL: NCT02337127
Title: A Prospective, Open-label, Multicenter Study of Lamivudine Extending Therapy in Chronic Hepatitis B Patients After 3-year of Oral Antiviral Agents
Brief Title: Lamivudine Extending Therapy in Chronic Hepatitis B Patients After 3-year of Oral Antiviral Agents
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUH-IRB-20110187
Record Dates: First submitted 2014-12-01; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): 250 treatment-naïve CHB patients who received at least 3-year of oral antiviral agents will receive Lamivudine extending therapy for 5 years.
  Interventions: Drug: Lamivudine
- Arm B (No Intervention): 250 treatment-naïve CHB patients who received at least 3-year of oral antiviral agents will receive follow-up.

INTERVENTIONS:
Drug: Lamivudine — Lamivudine, 100mg/day, per os
  Other Names: Zeffix
  Arms: Arm A

SUMMARY:
Current treatment guidelines indicate that oral antiviral agents for HBeAg-positive chronic hepatitis B virus infection (CHB) can be stopped if the patient has undergone HBeAg seroconversion with HBV-DNA loss measured at two consecutive occasions at least 6 months apart (primary treatment endpoint). Stopping treatment can be considered if undetectable HBV-DNA has been documented on three separate occasions 6 months apart in HBeAg-negative patients. However, oral antiviral drugs currently approved for the treatment of CHB have relatively limited sustained long-term efficacy and a large proportion of patients will suffer from HBV recurrence after stopping treatment.

DETAILED DESCRIPTION:
The purposes of this study are:

1. To evaluate the long-term efficacy of Lamivudine extending therapy in CHB patients who received at least 3-year of oral antiviral agents.
2. To evaluate the long-term outcomes and predictive factors of Lamivudine extending therapy in CHB patients who received at least 3-year of oral antiviral agents.

A prospective, open-label, multicenter study will enroll 500 treatment-naïve CHB patients who received at least 3-year of oral antiviral agents. With their voluntary decision after consultation, 250 patients will receive Lamivudine extending therapy for 5 years and the other 250 patients will receive follow-up and serve as controls. The primary outcome measurement is HBV DNA recurrence, whilst the secondary outcome measurement is liver-related outcomes and associated predictive factors

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients >=18 years of age
2. Negative serum HBV DNA within 3 months prior to entry
3. ALT <1.5 ULN within 3 months prior to entry
4. Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of test drug. Additionally, all fertile males with partners of childbearing age and females of the Lamivudine treatment arm must be using reliable contraception during the study and for 6 months after treatment completion.

Exclusion Criteria:

1. Women with ongoing pregnancy or breast feeding
2. Therapy with any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) *6 months prior to the first dose of study drug
3. Any investigational drug *6 weeks prior to the first dose of study drug
4. Co-infection with active hepatitis A, hepatitis C and/or human immunodeficiency virus (HIV)
5. Patients who have virological evidence of Lamivudine-associated YMDD mutants.
6. Patients who have clinical evidence of liver cirrhosis or hepatocellular carcinoma.
7. History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
8. Signs or symptoms of hepatocellular carcinoma
9. History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
10. Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening
11. Serum creatinine level >1.5 times the upper limit of normal at screening
12. History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
13. History of a severe seizure disorder or current anticonvulsant use
14. History of immunologically mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
15. Evidence of drug abuse (including excessive alcohol consumption) within one year of study entry
16. Inability or unwillingness to provide informed consent or abide by the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Rate of HBV DNA recurrence | up to 12 months

SECONDARY OUTCOMES:
Associated predictive factors of HBV DNA recurrence | up to 12 months
Rate of drug resistant mutation | up to 12 months
Rate of clinical relapse in Group B (non-intervention) | up to 12 months
  clinical relapse means HBV DNA>2000 IU/mL plus ALT > 2 fold upper limit of normal (ULN) in end of entecavir (ETV) normal alanine aminotransferase (ALT) or 2 fold elevation in end of ETV abnormal ALT patients

OTHER OUTCOMES:
Rate of severe reactivation or death | up to 12 months
  severe reactivation means alanine aminotransferase (ALT) > 10 fold upper limit of normal plus either total bilirubin > 2 mg/dL or prothrombin time prolong > 3 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Long Chuang, Principal Investigator — Kaohsiung Medical University Hospital, Internal Medicine
Locations (1):
- Hepatobiliary Division, Department of Internal Medicine, Kaohsiung Medical University Hospital, Kaohsiung City, NRW, Taiwan